CLINICAL TRIAL: NCT05444075
Title: A Method for Communication With Arabic Patients Suffering From Classic Locked- in Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Elnady, Professor of Neurology, Sohag University
Other Study IDs: Soh-Med-22-03-39
Record Dates: First submitted 2022-05-16; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Locked- in Syndrome
MeSH Terms: conditions — Coma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- subjects with preparatory education level: Ten subjects have a preparatory education level
  Interventions: Other: a method for communication
- subjects with high school education: ten subjects with a high school education or its equivalent
  Interventions: Other: a method for communication
- subjects with university education: ten subjects who have a university education, or are still in a university education stage
  Interventions: Other: a method for communication

INTERVENTIONS:
Other: a method for communication — the Arabic alphabet (arranged in the traditional order) printed on double-sided cardboard, with one copy facing the person and one facing the doctor.
  The code will be in the case of a positive selection (the desired line or letter) by looking up or one blink, but in the case of a negative selection (not the desired line or letter), it will be by looking down or two blinks.
  The person will choose the letters of each word and then choose the end of the word and after selecting all the words of the sentence choose the end of the sentence.
  After the strategy has been taught to the subject, he or she will be asked to communicate with the physician using this way.

SUMMARY:
Aim of the work The aim of this study is to test an Arabic alphabet communication system designed to train physicians to communicate with Arabic-speaking patients with LIS.

Subjects and methods

* Place of study: Department of Neurology at Sohag university hospital
* Type of study: clinical trial.
* Subjects: Thirty healthy subjects from three different educational levels. Ten subjects have a preparatory education level, ten subjects with a high school education or its equivalent, and ten subjects who have a university education or are still in a university education stage. They will be collected from among patients' relatives and employees of Sohag University Hospital.

Methods of the study: The method shown in the figure No. 1 is the Arabic alphabet (arranged in the traditional order) printed on double-sided cardboard, with one copy facing the person and one facing the doctor.

The code will be in the case of a positive selection (the desired line or letter) by looking up or one blink, but in the case of a negative selection (not the desired line or letter), it will be by looking down or two blinks.

The person will choose the letters of each word and then choose the end of the word and after selecting all the words of the sentence choose the end of the sentence.

After the strategy has been taught to the subject, he or she will be asked to communicate with the physician using this way.

DETAILED DESCRIPTION:
Aim of the work The aim of this study is to test an Arabic alphabet communication system designed to train physicians to communicate with Arabic-speaking patients with LIS.

Subjects and methods

* Place of study: Department of Neurology at Sohag university hospital
* Type of study: clinical trial.
* Subjects: Thirty healthy subjects from three different educational levels. Ten subjects have a preparatory education level, ten subjects with a high school education or its equivalent, and ten subjects who have a university education or are still in a university education stage. They will be collected from among patients' relatives and employees of Sohag University Hospital.

Methods of the study: the Arabic alphabet (arranged in the traditional order) printed on double-sided cardboard, with one copy facing the person and one facing the doctor.

The Arabic alphabet was divided into 4 groups and it was taken into account - as far as possible - to include letters of similar shape in the same group. Each group is listed on a separate line and given a number from 1 to 4 in addition to the letters, each line includes an option at the end of it to enable the person to change the line.

A fifth line has also been added that contains options for ending the word, ending the sentence, choosing numbers (which were included in a separate sixth line from 0 to 9) in addition to an option to change the line depends on the vertical eye movement or the blink of the eye lid and will be used in both ways.

The code will be in the case of a positive selection (the desired line or letter) by looking up or one blink, but in the case of a negative selection (not the desired line or letter), it will be by looking down or two blinks.

The person will choose the letters of each word and then choose the end of the word and after selecting all the words of the sentence choose the end of the sentence.

After the strategy has been taught to the subject, he or she will be asked to communicate with the physician using this way.

The researcher will present the subject a piece of paper on which is written all of the information that has to be communicated to the doctor. The researcher will notice that the method of communication was solely based on eye or eyelid movement, and if the person completes the communication in any other way (such as speech or head or hand movement), the attempt will be considered incorrect and will be repeated with a different piece of information.

For each person, at least four successful attempts with four different pieces of information will be made. Three of them will be information from the researcher to the person who will deliver it to the doctor, and the fourth will be a question from the doctor to the person who will then receive an answer from him.

A successful attempt is one that is made in the correct manner, regardless of whether the translated information is correct or incorrect.

All data will be collected, tabulated and statistically analyzed.

References Bauer, G., F. Gerstenbrand and E. Rumpl (1979). "Varieties of the locked-in syndrome." Journal of Neurology 221(2): 77-91.

Chisholm, N. and G. Gillett (2005). "The patient's journey: Living with locked-in syndrome." Bmj 331(7508): 94-97.

Khanna, K., A. Verma and B. Richard (2011). ""The locked-in syndrome": Can it be unlocked?" Journal of Clinical Gerontology and Geriatrics 2(4): 96-99.

Laureys, S., F. Pellas, P. Van Eeckhout, S. Ghorbel, C. Schnakers, F. Perrin, J. Berré, M.-E. Faymonville, K.-H. Pantke, F. Damas, M. Lamy, G. Moonen and S. Goldman (2005). The locked-in syndrome : what is it like to be conscious but paralyzed and voiceless? Progress in Brain Research. S. Laureys, Elsevier. 150: 495-611.

Smith, E. and M. Delargy (2005). "Locked-in syndrome." BMJ 330(7488): 406.

ELIGIBILITY:
Inclusion Criteria:

* educated healthy subjects

Exclusion Criteria:

* non-educated, healthy subjects
* subjects with any sensory deficits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty healthy subjects from three different educational levels. Ten subjects have a preparatory education level, ten subjects with a high school education or its equivalent, and ten subjects who have a university education or are still in a university education stage. They will be collected from among patients' relatives and employees of Sohag University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Alphabetic communication | up to 24 weeks
  The participant's ability to communicate in the Arabic alphabet using vertical eye movement